CLINICAL TRIAL: NCT02150473
Title: Delayed Gadolinium-enhanced Magnetic Resonance (MR) Imaging of Cartilage - A Pilot Study to Measure the Effect of Adalimumab Plus MTX Versus Placebo Plus MTX on Cartilage in Early RA Patients
Brief Title: The Effect of Adalimumab Plus Methotrexate (MTX) Versus Placebo Plus MTX on Cartilage in (RA) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAR-ERA; 2013-004604-19 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-05-29 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental): receive adalimumab 40 mg eow injections in combination with MTX for 24 weeks
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): receive placebo injections in combination with MTX for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — adalimumab 40 mg every other week in combination with MTX for 24 weeks
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebo — Placebo the same amount as adalimumab
  Arms: Placebo

SUMMARY:
This study aims to compare longitudinally the effect of adalimumab plus methotrexate (MTX) versus MTX monotherapy on cartilage GAG content, reflected by Delayed Gadolinium-enhanced magnetic resonance imaging of cartilage (dGEMRIC) index, in patients with early progressive rheumatoid arthritis (RA), who had not previously received any Disease modifying antirheumatic drug (DMARD) or biologic treatment.

DETAILED DESCRIPTION:
Patients will be randomly assigned to either adalimumab q2w plus oral MTX qw combination therapy or oral MTX qw monotherapy plus placebo subcutaneous (SC) q2w in a ration 2:1. To maintain blinding, matching placebo SC injections will be dispensed q2w to the MTX monotherapy group. All subjects will receive open-label MTX 15 mg qw as oral tablets. All subjects will take approximately 5 mg weekly dietary supplement of oral folate throughout the study on any day beginning 48 hours after ingestion of their oral study medication. Defined as standard therapy oral folate supplementation will be taken in a single dose 24-48 h after MTX therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of early RA (ERA) fulfilling the 2010 American college of rheumatology (ACR) criteria for classification of RA
* Disease duration less than 12 months from symptoms onset.

Exclusion Criteria:

* Subject has previous exposure to any systemic biologic therapy (e.g. abatacept, tocilizumab) including anti-Tumor necrosis factor (TNF therapy) (e.g., infliximab, golimumab, certolizumab pegol, etanercept) including adalimumab.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Joint space narrowing of the metacarpophalangeal (MCP II) and MCP III joints in the clinically dominant hand measured by variable flip-angle imaging 3 time (3T) MRI | 104 weeks
  Joint space narrowing will be measured by variable flip-angle imaging 3T MRI at week 24 and baseline. A possible reduction of the joint space narrowing should be seen by comparing mean intergroup difference of pooled (per patient) dGEMRIC index (T1 [ms]).

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Ostendorf, Prof.Dr., Principal Investigator — Poliklinik für Rheumatologie
Locations (1):
- Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany